CLINICAL TRIAL: NCT01577303
Title: Reduction of Social Phobia Symptoms With Internet-Based Cognitive Bias Modification
Brief Title: Treatment of Social Phobia With Cognitive Bias Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Attention training
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Social Phobia
Keywords: social phobia; social anxiety; cognitive bias modification
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- CBM training program variant 1 (Experimental): Attention training towards positive cues using words as stimuli
  Interventions: Behavioral: Cognitive bias modification training program variant 1
- CBM training program variant 2 (Experimental): Attention training towards positive cues using words and faces as stimuli
  Interventions: Behavioral: Cognitive bias modification training program variant 2
- CBM training program variant 3 (Experimental): Attention training towards negative using words as stimuli
  Interventions: Behavioral: CBM training program variant 3
- CBM training program variant 4 (Experimental): Attention training towards negative using words and faces
  Interventions: Behavioral: CBM training program variant 4
- Control training variant 1 (Experimental): Control training condition using words as stimuli
  Interventions: Behavioral: Control training variant 1
- Control training variant 2 (Experimental): Control training condition using words and faces as stimuli
  Interventions: Behavioral: Control training variant 2

INTERVENTIONS:
Behavioral: Cognitive bias modification training program variant 1 — Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 1. Participant is exposed to two words -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words and is then asked to press the corresponding arrow button on a keyboard. A total of 192 word pairs are shown during a session, of one third is the neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more positive word.
  Arms: CBM training program variant 1
Behavioral: Cognitive bias modification training program variant 2 — Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 2. Participant is exposed to a pair of words or a pair of faces -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words or faces and is then asked to press the corresponding arrow button on a keyboard. A total of 96 word pairs and 96 face pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more positive word or face.
  Arms: CBM training program variant 2
Behavioral: CBM training program variant 3 — Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 3. Participant is exposed to two words -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words and is then asked to press the corresponding arrow button on a keyboard. A total of 192 word pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more negative word.
  Arms: CBM training program variant 3
Behavioral: CBM training program variant 4 — Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 4. Participant is exposed to a pair of words or a pair of faces -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words or faces and is then asked to press the corresponding arrow button on a keyboard. A total of 96 word pairs and 96 face pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more negative word or face.
  Arms: CBM training program variant 4
Behavioral: Control training variant 1 — Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 1. Participant is exposed to a pair of words -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words and is then asked to press the corresponding arrow button on a keyboard. A total of 192 word pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe follows the more positive word and the more negative word with equal frequency..
  Arms: Control training variant 1
Behavioral: Control training variant 2 — Computerized, internet-based control training program, variant 2. Participant is exposed to a pair of words or a pair of faces -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words or faces and is then asked to press the corresponding arrow button on a keyboard. A total of 96 word pairs and 96 face pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe follows the more positive stimulus and the more negative stimulus with equal frequency.
  Arms: Control training variant 2

SUMMARY:
The purpose of this study is to determine whether different internet-based treatment programs, consisting of cognitive bias modification, reduce symptoms of social phobia among a population diagnosed with this disorder.

DETAILED DESCRIPTION:
Previous studies have shown that individuals with social phobia have attention biases, often focusing on aversive stimuli or avoiding aversive stimuli. Computerized training programs have been developed to implicitly direct the users attention towards a neutral, non-threatening stimuli. In this study, such a program will be provided to 128 participants that meet the diagnostic criteria for social phobia. It will be compared with a program that implicitly directs the users' attention towards threatening cues. Pre/post-measurements will be compared. Participants will be randomized to one of three groups, receiving one of the two variants of the cognitive bias modification program or a control training.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided
* Diagnosed social phobia (according to DSM-IV criteria)
* Access to computer with internet connection, and printer

Exclusion Criteria:

* Severe depression (and/or suicidal behavior)
* Addiction and/or abuse
* Suffer from other severe psychiatric condition (e.g. psychosis)
* Non-stable use of medication
* Undergoing other, parallel psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Liebowitz Social Anxiety Scale Self-Rated (LSAS-SR) | 24 hours
  The Liebowitz Social Anxiety Scale (LSAS) is a questionnaire by psychiatrist and researcher, Michael Liebowitz, whose objective is to assess the range of social interaction and performance situations which patients with social anxiety disorder may fear. It is commonly used to study outcomes in clinical trials. The scale features 24 items, 13 relating to performance anxiety and 11 concerning social situations. It is not intended for use as a self-reporting diagnosis.
Change from baseline in Liebowitz Social Anxiety Scale Self-Rated (LSAS-SR) | 14 days
  The Liebowitz Social Anxiety Scale (LSAS) is a questionnaire by psychiatrist and researcher, Michael Liebowitz, whose objective is to assess the range of social interaction and performance situations which patients with social anxiety disorder may fear. It is commonly used to study outcomes in clinical trials. The scale features 24 items, 13 relating to performance anxiety and 11 concerning social situations. It is not intended for use as a self-reporting diagnosis.
Change from baseline in Liebowitz Social Anxiety Scale Self-Rated (LSAS-SR) | 4 months
  The Liebowitz Social Anxiety Scale (LSAS) is a questionnaire by psychiatrist and researcher, Michael Liebowitz, whose objective is to assess the range of social interaction and performance situations which patients with social anxiety disorder may fear. It is commonly used to study outcomes in clinical trials. The scale features 24 items, 13 relating to performance anxiety and 11 concerning social situations. It is not intended for use as a self-reporting diagnosis.

SECONDARY OUTCOMES:
Change from baseline in Quality Of Life Inventory (QOLI) | 24 hours
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 14 days
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 4 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 24 hours
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 14 days
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 4 months
  9-item depression rating scale.
Change from baseline in Social Phobia Scale + Social Interaction Anxiety Scale | 24 hours
  Self-rated measurements of social anxiety/phobia.
Change from baseline in Social Phobia Scale + Social Interaction Anxiety Scale | 14 days
  Self-rated measurements of social anxiety/phobia.
Change from baseline in Social Phobia Scale + Social Interaction Anxiety Scale | 4 months
  Self-rated measurements of social anxiety/phobia.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Principal Investigator — Department of Psychology, Umeå University
Locations (1):
- Department of Psychology, Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Result] Boettcher J, Leek L, Matson L, Holmes EA, Browning M, MacLeod C, Andersson G, Carlbring P. Internet-based attention bias modification for social anxiety: a randomised controlled comparison of training towards negative and training towards positive cues. PLoS One. 2013 Sep 30;8(9):e71760. doi: 10.1371/journal.pone.0071760. eCollection 2013. PMID 24098630